CLINICAL TRIAL: NCT00245960
Title: A RANDOMIZED, OPEN-LABEL, TWO-PERIOD STUDY TO EVALUATE THE SAFETY AND EFFICACY OF ETANERCEPT ON SKIN AND JOINT DISEASE IN PSORIASIS SUBJECTS WITH PSORIATIC ARTHRITIS
Brief Title: Study Evaluating Etanercept on Skin and Joint Disease in Psoriatic Arthritis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0881A5-401; 2005-001533-15 (EudraCT Number); B1801271 (Other: Alias Study Number)
Record Dates: First submitted 2005-10-26; First posted 2005-10-28 (Estimated); Results first posted 2009-05-27 (Estimated); Last update posted 2022-01-31 (Actual); Status verified 2021-11

CONDITIONS: Psoriatic Arthritis
Keywords: Psoriatic Arthritis; Skin Disease; Joint Disease
MeSH Terms: conditions — Arthritis, Psoriatic; Skin Diseases; Joint Diseases | interventions — Etanercept

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator): Period 1 (Double Blind): 50mg bi-weekly (BIW) for weeks 1-12. Period 2 (Open Label): 50 mg weekly (QW).
  Interventions: Drug: etanercept
- B (Active Comparator): Period 1 (Double Blind): 50mg weekly (QW) with matching placebo for weeks 1-12. Period 2 (Open Label): 50 mg weekly (QW) for weeks 13-24.
  Interventions: Drug: etanercept; Drug: Placebo

INTERVENTIONS:
Drug: etanercept
  Arms: B
Drug: etanercept
  Arms: A
Drug: Placebo
  Arms: B

SUMMARY:
The purpose of the study was to compare the efficacy of 2 different Etanercept regimens for the treatment of skin and joint manifestations of psoriatic arthritis.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria:

* 18 years of age or older at time of consent
* Active Psoriatic Arthritis
* Clinically stable, plaque psoriasis involving more than 10% of the body surface area

Exclusion Criteria:

Exclusion Criteria:

* Evidence of skin conditions other than psoriasis that would interfere with skin examinations.
* Systemic anti-psoriasis therapy or DMARD within 28 days of study drug initiation
* Prior exposure to any TNF-inhibitor, including etanercept

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 752 (Actual)
Dates: Start 2005-12-27 (Actual); Primary Completion 2008-03-29 (Actual); Study Completion 2008-03-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (114):
- Argentina (5):
  - Hospital A Posadas, Palomar, Buenos Aires
  - Hospital General de Agudos, Buenos Aires
  - Hospital Italiano de Buenos Aires, Buenos Aires
  - CEMIC, Buenos Aires
  - Instituto de Medicina Cutanea, Buenos Aires
- Australia (2):
  - Goulburn Street Medical Centre, Liverpool, New South Wales
  - St Vincent's Hospital VIC, Fitzroy
- Austria (2):
  - Universitaetsklinik Graz, Graz, SM
  - Krankenhaus Rudolfsstiftung, Vienna
- Belgium (2):
  - Universitair Ziekenhuis Gent, Ghent
  - CHU Liege, Liège
- Colombia (2):
  - Centro Integral de Reumatologia del Caribe S.A.S, Barranquilla, Atlántico
  - Centro Medico de la Sabana, Bogotá
- Czechia (3):
  - Centrum Rehabilitace, Zlín, Czech Republic
  - Revmatologicky ustav, Prague
  - Revmatologicka Ambulance, Uherské Hradiště
- Denmark (5):
  - Bispebjerg University Hospital, Copenhagen
  - Gentofte University Hospital, Hellerup
  - Hørsholm hospital, Hørsholm
  - Odense University Hospital, Odense C
  - University of Copenhagen - Roskilde Hospital, Roskilde
- Finland (3):
  - Mehiläinen Terveyspalvelut Oy Forum, Helsinki
  - Tampereen Reumatoismisto, Tampere
  - Iho ja Allergiapulssi, Turku
- France (13):
  - Centre Hospitalier du Mans, Le Mans, Cedex
  - Hôpital Saint André, Bordeaux
  - CHU - Hôpital Morvan, Brest
  - C.H.R.U. de Caen, Caen
  - Hôpital Henri Mondor, Créteil
  - CHU Dupuytren, Limoges
  - CHU de l Archet, Nice
  - Hopital Saint Louis, Paris
  - Hôpital Bichat - Claude Bernard, Paris
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - CHU La Milétrie, Poitiers
  - CHU - Hopital Charles Nicolle, Rouen
  - CHRU- Hôpital Trousseau, Tours
- Germany (18):
  - Fachklinik Bad Bentheim, Bad Bentheim
  - Klinik fuer Dermatologie, Venerologie und Allergologie, Berlin
  - Schonhauser Allee 71, Berlin
  - Hautarztpraxis Dr. Margrit Simon, Berlin
  - Klinische Forschung Berlin-Buch GmbH, Berlin
  - Schlossparkklinik Berlin, Berlin
  - Klinik und Poliklinik für Dermatologie der Friedrich-Wilhelm, Bonn
  - Allgemeines Krankenhaus Eilbek, Eilbek
  - Universitätsklinikum Hartmmannstrasse 14 Erlangen 91052, Erlangen
  - Klinikum der J.W. Goethe-Universitat, Frankfurt
  - Georg-August Universitaet Goettingen, Göttingen
  - SCIderm GmbH Hamburg, Hamburg
  - Friedrich-Schiller Universitat Jena, Jena
  - Bahnhofstr. 1, Mahlow
  - Klinikum Innenstadt der Universitaet Muenchen, München
  - Dermatologische Gemeinschaftspraxis Rosenbach, Osnabrück
  - Praxis Dr. M. Richter, Rostock
  - Universitaetsklinik Wuerzburg, Würzburg
- University of Athens Andreas Syngros Hospital Athens, Greece, Athens, Greece
- Hungary (6):
  - Semmelweis University - Faculty of Health Sciences, Budapest
  - Debreceni Egyetem Orvos és Egészségtudományi Centrum, Debrecen
  - Miskolc Megyei Jogu Varos Onkormanyzata, Miskolci Egeszsegui, Miskolc
  - Pecsi Tudomanyegyetem, AOK, Pécs
  - Medical University of Szeged, Szeged
  - HETENYI Geza Hospital, Szolnok
- Italy (8):
  - Azienda Ospedaliera Spedali Civili di Brescia, Brescia
  - Ospedale San Giovanni di Dio, Cagliari
  - Clinica Dermatologica, Catania
  - Ospedale Galeazzi, Milan
  - Universita degli Studi di Parma, Parma
  - Policlinico Umberto I - Universita La Sapienza, Roma
  - Idi-Irccs, Roma
  - Universita degli Studi di Siena, Siena
- Mexico (2):
  - Unidad de Investigacion en, Guadalajara, Jalisco
  - CLIDITER S.A. de C.V., Mexico City
- Netherlands (5):
  - University Medical Center St. Radboud, Nijmegen, GA
  - Academisch Ziekenhuis Maastricht, Maastricht, THE Netherlands
  - Ziekenhuis Walcheren, Flushing
  - Academisch Ziekenhuis Maastricht, Maastricht
  - Diaconessenhuis Voorburg, Voorburg
- Poland (4):
  - Akad. Medyczna im L. Rydygiera, Bydgoszcz
  - Samodzielny Publiczny Szpital Kliniczny nr 4, Lublin
  - Wojskowy Instytut Medyczny, Warsaw
  - Zesp. Naukowo-Kliniczny IWOLANG, Uzdrowiskowa Klinika Dermat, Warsaw
- Portugal (2):
  - Hospitais Da Universidade De Coimbra, Coimbra
  - Hospital Santo Antonio, Porto
- King Faisal Specialist Hospital & Research Centre, Riyadh, Saudi Arabia
- Serbia and Montenegro (4):
  - Institute of Rheumatology Belgrade, Belgrade
  - Institute of Rheumatology Niska Banja, Niska Banja
  - Clinic for Dermatology and Clinic for Medical Rehabilitation, Novi Sad
  - Clinical Center Zemun, Zemun
- South Korea (2):
  - Seoul National University Hospital, Seoul
  - Asan Medical Centre, Seoul
- Spain (7):
  - Hospital Universitario Puerto Real, Puerto Real, Cadiz
  - Hospital de Donostia, San Sebastián, Guipúzcua
  - Hospital Insular de Canarias, Las Palmas de Gran Canaria, Isalas Canarias
  - Hospital Severo Ochoa de Leganes, Leganés, Madrid
  - Hospital Nuestra Senora Del Mar, Barcelona
  - Hospital de la Santa Cruz y San Pablo, Barcelona
  - Hospital Ramon y Cajal, Madrid
- Sweden (3):
  - Länssjukhuset Ryhov, Jönköping
  - Umeå University Hospital, Umeå
  - Akademiska Sjukhuset i Uppsala, Uppsala
- Switzerland (2):
  - CHUV Lausanne, Lausanne
  - Universitatsspital Zurich, Zurich
- Taiwan (2):
  - Chang Gung Memorial Hospital-Kaohsiung, Kaohsiung Hsiang, Taiwan, R.o.c.
  - National Taiwan University Hospital, Taipei TOC
- Hacettepe University Medicine Faculty, Ankara, Turkey (Türkiye)
- United Kingdom (9):
  - The Royal Free Hospital, Pond Street, Hampstead, London, Hampstead
  - Hope Hospital, Salford, Lancashire
  - Harrogate District Hospital, Harrogate, North Yorkshire
  - Leeds General Infirmary, Leeds, Leeds, Yorkshire
  - Aberdeen Royal Infirmary, Aberdeen
  - University Hospital of Wales, Cardiff
  - The Royal Free Hospital, Pond Street, Hampstead, London
  - Guy's and St. Thomas' Trust St.Thomas' Hospital, London
  - George Elliott Hospital, Nuneaton

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Coates LC, Gottlieb AB, Merola JF, Boone C, Szumski A, Chhabra A. Comparison of Different Remission and Low Disease Definitions in Psoriatic Arthritis and Evaluation of Their Prognostic Value. J Rheumatol. 2019 Feb;46(2):160-165. doi: 10.3899/jrheum.180249. Epub 2018 Oct 15. PMID 30323006
- [Derived] Griffiths CE, Christophers E, Szumski A, Jones H, Mallbris L. Impact of early vs. late disease onset on treatment response to etanercept in patients with psoriasis. Br J Dermatol. 2015 Nov;173(5):1271-3. doi: 10.1111/bjd.13865. Epub 2015 Aug 17. No abstract available. PMID 25913550
- [Derived] Kirkham B, de Vlam K, Li W, Boggs R, Mallbris L, Nab HW, Tarallo M. Early treatment of psoriatic arthritis is associated with improved patient-reported outcomes: findings from the etanercept PRESTA trial. Clin Exp Rheumatol. 2015 Jan-Feb;33(1):11-9. Epub 2014 Dec 22. PMID 25535650
- [Derived] Griffiths CE, Sterry W, Brock F, Dilleen M, Stefanidis D, Germain JM, Mallbris L. Pattern of response in patients with moderate-to-severe psoriasis treated with etanercept. Br J Dermatol. 2015 Jan;172(1):230-8. doi: 10.1111/bjd.13139. Epub 2014 Nov 13. PMID 24861696
- [Derived] Gniadecki R, Robertson D, Molta CT, Freundlich B, Pedersen R, Li W, Boggs R, Zbrozek AS. Self-reported health outcomes in patients with psoriasis and psoriatic arthritis randomized to two etanercept regimens. J Eur Acad Dermatol Venereol. 2012 Nov;26(11):1436-43. doi: 10.1111/j.1468-3083.2011.04308.x. Epub 2011 Oct 31. PMID 22035157
- [Derived] Sterry W, Ortonne JP, Kirkham B, Brocq O, Robertson D, Pedersen RD, Estojak J, Molta CT, Freundlich B. Comparison of two etanercept regimens for treatment of psoriasis and psoriatic arthritis: PRESTA randomised double blind multicentre trial. BMJ. 2010 Feb 2;340:c147. doi: 10.1136/bmj.c147. PMID 20124563
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=0881A5-401&StudyName=Study%20evaluating%20Etanercept%20on%20Skin%20and%20Joint%20Disease%20in%20Psoriatic%20Arthritis

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited worldwide from December 2005 to September 2007.
Pre-assignment Details: Subjects were screened up to 4 weeks.
Groups:
- Etanercept BIW/QW: Period 1 (Double blind): etanercept 50mg bi-weekly (BIW) for weeks 1-12. Period 2 (Open Label): etanercept 50mg weekly (QW) for weeks 13-24.
- Etanercept QW/QW: Period 1 (Double blind): etanercept 50mg weekly (QW) with matching placebo for weeks 1-12. Period 2 (Open Label): etanercept 50mg weekly (QW) for weeks 13-24.
Period: Period 1 (Double Blind): 1-12 Weeks
Arm/Group | Etanercept BIW/QW | Etanercept QW/QW
Started | 379 | 373
Completed | 364 | 362
Not Completed | 15 | 11
Not completed — Adverse Event | 6 | 7
Not completed — Pregnancy | 0 | 1
Not completed — Withdrawal of consent | 2 | 0
Not completed — Unsatisfactory Response | 2 | 1
Not completed — Protocol Violation | 3 | 0
Not completed — Withdrawal by Subject | 2 | 2
Period: Period 2 (Open Label): 13-24 Weeks
Arm/Group | Etanercept BIW/QW | Etanercept QW/QW
Started | 364 | 362
Completed | 350 | 344
Not Completed | 14 | 18
Not completed — Adverse Event | 8 | 4
Not completed — Lost to Follow-up | 2 | 2
Not completed — Unsatisfactory Response | 2 | 5
Not completed — Withdrawal by Subject | 1 | 3
Not completed — Protocol Violation | 1 | 3
Not completed — Withdrawal of consent | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Etanercept BIW/QW | Etanercept QW/QW | Total
Number analyzed (Participants) | 379 | 373 | 752
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.11 (11.39) | 46.93 (11.41) | 46.52 (11.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 136 | 143 | 279
  Male | 243 | 230 | 473

OUTCOME MEASURES:

1. Secondary Outcome: Number of Patients Achieving Psoriatic Arthritis Response Criteria (PsARC)
Description: The PsARC response was defined as improvement in at least 2 of the four criteria: >=30% decrease in swollen joint count, >=30% decrease in tender joint count, >=20% improvement in patient's Global Assessment of Disease Activity (arthritis) using VAS (0-100 mm, 0=excellent and 100= poor), >=20% improvement in physician's Global Assessment of Disease Activity using VAS (VAS: 0-100 mm, 0=no arthritis activity and 100=extremely active arthritis), and at least one of the 2 joint criteria with no deterioration in the other criteria.
Time Frame: 12 and 24 weeks
Population: The analysis population was the Modified Intent to Treat (mITT) population which includes all randomized patients who received ≥ 1 dose of study drug and had at least 1 post baseline efficacy evaluation. Last observation carried forward (LOCF) approach used for missing data imputation.
Measure: Number; unit: participants
Arm/Group | Etanercept BIW/QW | Etanercept QW/QW
Number analyzed (Participants) | 372 | 372
participants
  At 12 Weeks: number analyzed (Participants) | 371 | 371
  At 12 Weeks | 284 | 282
  At 24 Weeks | 303 | 299

2. Primary Outcome: Number of Patients Achieving "Clear" or "Almost Clear" on Physician Global Assessment (PGA) of Psoriasis
Description: The PGA of Psoriasis scale ranges from 0 (no psoriasis) to 5 (severe disease). "Clear" and "Almost Clear" includes all patients who were scored as a 0 or 1.
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Etanercept BIW/QW | Etanercept QW/QW
Number analyzed (Participants) | 379 | 373
participants | 176 | 119

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Etanercept BIW/QW | Etanercept QW/QW
Serious Adverse Events (participants affected / at risk) | 15 | 11
Other Adverse Events (participants affected / at risk) | 213 | 190
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Etanercept BIW/QW | Etanercept QW/QW
Abdominal pain (General disorders) | 1/379 | 0/373
Abscess (General disorders) | 0/379 | 1/373
Accidental injury (General disorders) | 1/379 | 1/373
Fever (General disorders) | 1/379 | 0/373
Infection (Infections and infestations) | 1/379 | 2/373
Cerebral ischemia (Vascular disorders) | 1/379 | 1/373
Cerebrovascular accident (Vascular disorders) | 1/379 | 1/373
Myocardial ischemia (Cardiac disorders) | 1/379 | 0/373
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 0/379 | 1/373
Large intestine perforation (Gastrointestinal disorders) | 1/379 | 0/373
Melena (Gastrointestinal disorders) | 0/379 | 1/373
Nausea (Gastrointestinal disorders) | 1/379 | 0/373
Stomach ulcer hemorrhage (Gastrointestinal disorders) | 0/379 | 1/373
Vomiting (Gastrointestinal disorders) | 1/379 | 1/373
Anemia (Blood and lymphatic system disorders) | 1/379 | 0/373
Abnormal gait (Nervous system disorders) | 1/379 | 0/373
Depression (Nervous system disorders) | 1/379 | 0/373
Dizziness (Nervous system disorders) | 1/379 | 0/373
Paresthesia (Nervous system disorders) | 1/379 | 0/373
Chronic obstructive airways disease (Respiratory, thoracic and mediastinal disorders) | 1/379 | 0/373
Psoriasis (Skin and subcutaneous tissue disorders) | 2/379 | 1/373
Skin carcinoma (Skin and subcutaneous tissue disorders) | 2/379 | 1/373
Breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/379 | 0/373
Kidney pain (Renal and urinary disorders) | 0/379 | 1/373
Local reaction to procedure (General disorders) | 1/379 | 0/373
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | Etanercept BIW/QW | Etanercept QW/QW
Headache (General disorders) | 19/379 | 19/373
Injection site (General disorders) | 32/379 | 23/373
Cardiovascular general disorders (Cardiac disorders) | 24/379 | 23/373
Digestive general disorders (Gastrointestinal disorders) | 38/379 | 37/373
Metabolic and nutritional general disorders (Metabolism and nutrition disorders) | 23/379 | 20/373
Nervous general disorders (Nervous system disorders) | 24/379 | 18/373
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 22/379 | 24/373
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 50/379 | 36/373
Skin and appendages general disorders (Skin and subcutaneous tissue disorders) | 45/379 | 41/373

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.